CLINICAL TRIAL: NCT05151536
Title: To Explore the Impact of Epinephrine on Biomarkers of Nervous System Ischemia-reperfusion Injury in Patients With Stanford Type A Dissection
Brief Title: Effects of Different Doses of Epinephrine on Biomarkers of Nervous System Ischemia-reperfusion Injury in Patients With Stanford Type A Dissection
Status: Completed | Type: Observational
Sponsor: Yunlong Fan (Other)
Responsible Party: Sponsor-Investigator, Yunlong Fan, Clinical Professor, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: chinaPLAGH-66936749
Record Dates: First submitted 2021-11-28; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Adrenaline; Aortic Dissection; Drug Dose; Nervous System; Ischemia Reperfusion Injury
MeSH Terms: conditions — Aortic Dissection; Neurologic Manifestations; Reperfusion Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aortic dissection is the most common aortic disease leading to death. Among them, patients with Stanford type A dissection (TAAD) are prone to dissection rupture in the early stage, and their condition deteriorates rapidly. They need immediate surgical treatment after admission.In this study, the detection data of biomarkers of nervous system Ischemia / Reperfusion (I/R)injury in patients with Stanford type A dissection were retrospectively analyzed, and the effects of different doses of adrenaline on biomarkers of nervous system I/R injury were evaluated by statistical methods.The information of 132 patients with Stanford type A aortic dissection who underwent sun's operation in the Department of cardiovascular surgery of the first medical center of the PLA General Hospital from January 2012 to January 2019 was retrospectively analyzed.

ELIGIBILITY:
Inclusion Criteria:

* The patient's age was 18-75 years old; TAAD was diagnosed by aortic CTA before operation; Sun's operation was performed within two weeks of onset; Deep hypothermic circulatory arrest (DHCA) and selective unilateral cerebral perfusion via right axillary artery were used for brain protection; Adrenaline was used after operation

Exclusion Criteria:

* Nervous system disease and mental system disease before operation; Recent acute coronary syndrome; Recent cardiac arrest; Recent poor perfusion of visceral or peripheral organs; Recent hypoxemia; Previous history of cardiac surgery; Intraoperative death and death within 48 hours after operation; Neurological or psychiatric symptoms occurred within 48 hours after operation; Adrenaline was not used after operation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The TAAD patients aged 18-75 years old
Sampling Method: Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Biomarkers of nervous system ischemia-reperfusion injury | 24 hours
  Monoamine oxidase, superoxide dismutase, interleukin-6, tumor necrosis factor- α

IPD SHARING:
Plan to Share IPD: Undecided